CLINICAL TRIAL: NCT06073561
Title: Underwater Endoscopic Mucosal Resection a Learning Curve Study
Brief Title: Underwater Endoscopic Mucosal Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Portugues Oncologia de Lisboa Francisco Gentil (Other)
Responsible Party: Principal Investigator, Luís Correia Gomes, Medical Degree, Instituto Portugues Oncologia de Lisboa Francisco Gentil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UIC/1593
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Colon Polyp; Adenoma Colon
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Every patient will be selected do underwater emr group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Underwater mucosectomy (Experimental): Every colonoscopy should be performed with a high definition colonoscope, such as Olympus series Q185 or Q190 with virtual chromoendoscopy by NBI (Olympus Inc., Tokyo, Japan) or Fujifilm EC-760R-V/L or EC-760Z-V/L with virtual chromoendoscopy by LBI (Fujifilm Group, Japan).
  A study investigator or a senior endoscopy fellow under their direct supervision should perform all procedures.
  The U-EMR procedure should include the following steps: CO2 should be completely removed, and the bowel lumen filled with normal saline using a water jet pump (OFP-2, Olympus Medical System or similar) until the lesion is totally immersed in water. The lesion and 2-3 mm of normal surrounding mucosa should be resected using electrocauterization (VIO 200D Endocut Q Effect 3; ERBE Electromedizin, Tübingen, Germany).
  Interventions: Other: learning curve of Underwater mucosectomy

INTERVENTIONS:
Other: learning curve of Underwater mucosectomy — Patients will be submitted to underwater mucosectomy (U-EMR)

SUMMARY:
The global aim of this multi-centric study is to assess the learning curve of U-EMR by an endoscopist skilled in C-EMR aiming to assess the application in real world and check the rate of complete EMR and adverse events related to the procedure.

DETAILED DESCRIPTION:
Conventional Endoscopic mucosal resection (C-EMR) is currently the standard therapy for the removal of large colon polyps. The procedure consists on the injection of fluids into the submucosa layer below the lesion with the intention to create a cushion to separate it from the muscular layer and avoid its damage and consequently perforation and thermal injury. There are some drawbacks about this technique such us fibrotic polyps, difficult location (areas behind the fold and appendicular orifice) and recurrence rate which without ablation techniques could reach 30%.

Underwater endoscopic mucosal resection (U-EMR) has been first described in 2012 by Binmoeller et al [10] and the main difference to C-EMR was the absence of need the submucosal injection. This would be possible because when the lumen is filled with water, the mucosal and the submucosal layer tend to float while the muscularis propria maintains its circular shape even in the presence of peristalsis. Recent data as shown not only a lower rate of recurrence but also a lower procedure time and R0 resections with no difference in adverse events.

Therefore, the global aim of this multi-centric study is to assess the learning curve of U-EMR by an endoscopist skilled in C-EMR aiming to assess the application in real world and check the rate of complete EMR and adverse events related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years-old or older with at least one large (>10 and <30 mm) non pedunculated polyp
* Agreement with study's procedures, having signed the informed consent for the study and EMR, prior to the procedure

Exclusion Criteria:

* Previous attempted resection
* Lesion located at ileo-cecal valve or appendiceal orifice
* Fully circumferential lesion
* Pedunculated polyps (Paris classification type Ip) and ulcerated depression lesions (Paris classification type III)
* Surface pattern suggestive of deep invasion (ex: narrow-band imaging (NBI) International Colorectal Endoscopic (NICE) classification type 3 criteria, Kudo V or equivalent)
* Invasive cancer at EMR specimen
* Inflammatory bowel disease
* Familial polyposis syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
learning curve of the application of U-EMR by endoscopists skilled in C-EMR | 6 months
  evaluate the learning curve of the application of U-EMR by endoscopists skilled in C-EMR after an online course about U-EMR technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No